CLINICAL TRIAL: NCT05635201
Title: Effects of Changes in Autonomic Nervous Activity on Changes in Blood Pressure After Anesthesia Induction: Remimazolam Versus Propofol
Brief Title: Changes in Autonomic Nervous Activity and Blood Pressure After Anesthesia Induction: Remimazolam Versus Propofol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daegu Catholic University Medical Center (Other)
Collaborators: Hana Pharm Co., Ltd. (Industry)
Responsible Party: Principal Investigator, JongHae Kim, Professor, Daegu Catholic University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CR-22-138
Record Dates: First submitted 2022-11-23; First posted 2022-12-02 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: General Anesthetics
MeSH Terms: interventions — Propofol; remimazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol group (Active Comparator): Receives propofol for anesthesia induction
  Interventions: Drug: Anesthesia induction with propofol
- Remimazolam group (Experimental): Receives remimazolam for anesthesia induction
  Interventions: Drug: Anesthesia induction with remimazolam

INTERVENTIONS:
Drug: Anesthesia induction with propofol — After a 10-minute-long acclimation, general anesthesia is induced with 2% propofol at the effect-site concentration of 4 μg/ml based on the Marsh Pharmacokinetic model. The effect-site concentration was maintained at 4 μg/ml until the trachea was intubated. Five minutes after the anesthesia induction, remifentanil was administered at the effect-site concentration of 4 ng/ml based on the Minto pharmacokinetic model until the trachea was intubated. With the initiation of remifentanil infusion, 1 mg/kg of rocuronium was administered following the calibration of the neuromuscular monitoring device. With the train-of-four count of 0, the trachea was intubated. Then, the effect-site concentrations of propofol and remifentanil were decreased to 3 μg/ml and 0 ng/ml, respectively, until the surgical incision was made.
  Arms: Propofol group
Drug: Anesthesia induction with remimazolam — After a 10-minute-long acclimation, general anesthesia is induced with a 2-minute-long infusion of remimazolam at a rate of 12 mg/kg/hr, after which the infusion rate was reduced to 1 mg/kg/hr and was maintained until the surgical incision was made. Five minutes after the anesthesia induction, remifentanil was administered at the effect-site concentration of 4 ng/ml based on the Minto pharmacokinetic model until the trachea was intubated. With the initiation of remifentanil infusion, 1 mg/kg of rocuronium was administered following the calibration of the neuromuscular monitoring device. With the train-of-four count of 0, the trachea was intubated. Then, the effect-site concentration of remifentanil was decreased to 0 ng/ml until the surgical incision was made.
  Arms: Remimazolam group

SUMMARY:
The goal of this clinical trial is to compare the effects of changes in autonomic nervous activity on changes in blood pressure after anesthesia induction between propofol and remimazolam in patients undergoing low-risk surgery. The main questions it aims to answer are:

* Does remimazolam shift sympathovagal balance toward parasympathetic predominance less than propofol?
* Does the less shift in sympathovagal balance toward parasympathetic predominance attenuate the reduction in blood pressure? Participants will be administered either propofol or remimazolam for anesthesia induction, after which the autonomic nervous activity and blood pressure will be measured.

Researchers will compare the propofol and remimazolam groups to see if remimazolam causes less shift in sympathovagal balance toward parasympathetic predominance and subsequently attenuates the reduction in blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 60 years
* American Society of Anesthesiologists physical status of 1
* Elective low-risk surgery requiring general anesthesia, the duration of which is shorter than 2 hours and 30 minutes (e.g., Laparoscopic cholecystectomy, Functional endoscopic sinus surgery, etc.)
* Body mass index less than 30 kg/m2

Exclusion Criteria:

* Arrhythmias or cardiac conduction disorders
* Disease or medical conditions affecting autonomic nervous activity (hypertension, diabetes mellitus, ischemic heart disease, congestive heart failure, cerebrovascular accident, chronic kidney disease, thyroid dysfunction, etc.)
* Valvular heart disease
* Use of medications affecting autonomic nervous activity or cardiac conduction (e.g., beta blocker)
* Limited mouth opening, limited head and upper neck extension, history of obstructive sleep apnea, or Modified Mallampati class 3 or 4
* Serum electrolyte abnormalities
* Severe hypovolemia
* Psychiatric diseases

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Difference in low-to-high frequency power ratio (LF/HF) of heart rate variability (HRV) between 5-minute-pre-anesthesia and 5-minute-post-anesthesia induction | Between 5 minutes before and after anesthesia induction
  Low-frequency power (LF) and high-frequency power (HF) of heart rate variability (HRV) were calculated with the Fast Fourier Transform applied to a 5-minute-long electrocardiogram (ECG) waveform. LF/HF represents the sympathovagal balance.

SECONDARY OUTCOMES:
Low-frequency power (LF) of heart rate variability (HRV) during 5 minutes before anesthesia induction | 5 minutes before anesthesia induction
  Low-frequency power (LF) of heart rate variability (HRV) were calculated by integrating power spectra between 0.04 and 0.15 Hz, which were obtained from the Fast Fourier Transform applied to a 5-minute-long electrocardiogram (ECG) waveform. LF represents the combined sympathetic and parasympathetic modulation of heart rate via baroreceptor reflexes, but is mainly modulated by sympathetic nervous activity.
Low-frequency power (LF) of heart rate variability (HRV) during 5 minutes after anesthesia induction | 5 minutes after anesthesia induction
  Low-frequency power (LF) of heart rate variability (HRV) were calculated by integrating power spectra between 0.04 and 0.15 Hz, which were obtained from the Fast Fourier Transform applied to a 5-minute-long electrocardiogram (ECG) waveform. LF represents the combined sympathetic and parasympathetic modulation of heart rate via baroreceptor reflexes, but is mainly modulated by sympathetic nervous activity.
Low-frequency power (LF) of heart rate variability (HRV) during 5 minutes after endotracheal intubation | 5 minutes after endotracheal intubation
  Low-frequency power (LF) of heart rate variability (HRV) were calculated by integrating power spectra between 0.04 and 0.15 Hz, which were obtained from the Fast Fourier Transform applied to a 5-minute-long electrocardiogram (ECG) waveform. LF represents the combined sympathetic and parasympathetic modulation of heart rate via baroreceptor reflexes, but is mainly modulated by sympathetic nervous activity.
Low-frequency power (LF) of heart rate variability (HRV) during 5 minutes before surgical incision | 5 minutes before surgical incision
  Low-frequency power (LF) of heart rate variability (HRV) were calculated by integrating power spectra between 0.04 and 0.15 Hz, which were obtained from the Fast Fourier Transform applied to a 5-minute-long electrocardiogram (ECG) waveform. LF represents the combined sympathetic and parasympathetic modulation of heart rate via baroreceptor reflexes, but is mainly modulated by sympathetic nervous activity.
High-frequency power (HF) of heart rate variability (HRV) during 5 minutes before anesthesia induction | 5 minutes before anesthesia induction
  High-frequency power (HF) of heart rate variability (HRV) were calculated by integrating power spectra between 0.15 and 0.4 Hz, which were obtained from the Fast Fourier Transform applied to a 5-minute-long electrocardiogram (ECG) waveform. HF represents the parasympathetic modulation of heart rate in response to respiration.
High-frequency power (HF) of heart rate variability (HRV) during 5 minutes after anesthesia induction | 5 minutes after anesthesia induction
  High-frequency power (HF) of heart rate variability (HRV) were calculated by integrating power spectra between 0.15 and 0.4 Hz, which were obtained from the Fast Fourier Transform applied to a 5-minute-long electrocardiogram (ECG) waveform. HF represents the parasympathetic modulation of heart rate in response to respiration.
High-frequency power (HF) of heart rate variability (HRV) during 5 minutes after endotracheal intubation | 5 minutes after endotracheal intubation
  High-frequency power (HF) of heart rate variability (HRV) were calculated by integrating power spectra between 0.15 and 0.4 Hz, which were obtained from the Fast Fourier Transform applied to a 5-minute-long electrocardiogram (ECG) waveform. HF represents the parasympathetic modulation of heart rate in response to respiration.
High-frequency power (HF) of heart rate variability (HRV) during 5 minutes before surgical incision | 5 minutes before surgical incision
  High-frequency power (HF) of heart rate variability (HRV) were calculated by integrating power spectra between 0.15 and 0.4 Hz, which were obtained from the Fast Fourier Transform applied to a 5-minute-long electrocardiogram (ECG) waveform. HF represents the parasympathetic modulation of heart rate in response to respiration.
Total power (TP) of heart rate variability (HRV) during 5 minutes before anesthesia induction | 5 minutes before anesthesia induction
  Total power (TP) of heart rate variability (HRV) were calculated by integrating power spectra between 0 and 0.4 Hz, which were obtained from the Fast Fourier Transform applied to a 5-minute-long electrocardiogram (ECG) waveform. TP represents the overall activity of the autonomic nervous system.
Total power (TP) of heart rate variability (HRV) during 5 minutes after anesthesia induction | 5 minutes after anesthesia induction
  Total power (TP) of heart rate variability (HRV) were calculated by integrating power spectra between 0 and 0.4 Hz, which were obtained from the Fast Fourier Transform applied to a 5-minute-long electrocardiogram (ECG) waveform. TP represents the overall activity of the autonomic nervous system.
Total power (TP) of heart rate variability (HRV) during 5 minutes after endotracheal intubation | 5 minutes after endotracheal intubation
  Total power (TP) of heart rate variability (HRV) were calculated by integrating power spectra between 0 and 0.4 Hz, which were obtained from the Fast Fourier Transform applied to a 5-minute-long electrocardiogram (ECG) waveform. TP represents the overall activity of the autonomic nervous system.
Total power (TP) of heart rate variability (HRV) during 5 minutes before surgical incision | 5 minutes before surgical incision
  Total power (TP) of heart rate variability (HRV) were calculated by integrating power spectra between 0 and 0.4 Hz, which were obtained from the Fast Fourier Transform applied to a 5-minute-long electrocardiogram (ECG) waveform. TP represents the overall activity of the autonomic nervous system.
Low-to-high-frequency power ratio (LF/HF) of heart rate variability (HRV) during 5 minutes before anesthesia induction | 5 minutes before anesthesia induction
  Low-frequency power (LF) and high-frequency power (HF) of heart rate variability (HRV) were calculated with the Fast Fourier Transform applied to a 5-minute-long electrocardiogram (ECG) waveform. LF/HF represents the sympathovagal balance.
Low-to-high-frequency power ratio (LF/HF) of heart rate variability (HRV) during 5 minutes after anesthesia induction | 5 minutes after anesthesia induction
  Low-frequency power (LF) and high-frequency power (HF) of heart rate variability (HRV) were calculated with the Fast Fourier Transform applied to a 5-minute-long electrocardiogram (ECG) waveform. LF/HF represents the sympathovagal balance.
Low-to-high-frequency power ratio (LF/HF) of heart rate variability (HRV) during 5 minutes after endotracheal intubation | 5 minutes after endotracheal intubation
  Low-frequency power (LF) and high-frequency power (HF) of heart rate variability (HRV) were calculated with the Fast Fourier Transform applied to a 5-minute-long electrocardiogram (ECG) waveform. LF/HF represents the sympathovagal balance.
Low-to-high-frequency power ratio (LF/HF) of heart rate variability (HRV) during 5 minutes before surgical incision | 5 minutes before surgical incision
  Low-frequency power (LF) and high-frequency power (HF) of heart rate variability (HRV) were calculated with the Fast Fourier Transform applied to a 5-minute-long electrocardiogram (ECG) waveform. LF/HF represents the sympathovagal balance.
Root mean square of the successive differences of the RR intervals (RMSSD) during 5 minutes before anesthesia induction | 5 minutes before anesthesia induction
  RMSSD represents the parasympathetic nervous activity mediated by a respiratory sinus arrhythmia.
Root mean square of the successive differences of the RR intervals (RMSSD) during 5 minutes after anesthesia induction | 5 minutes after anesthesia induction
  RMSSD represents the parasympathetic nervous activity mediated by a respiratory sinus arrhythmia.
Root mean square of the successive differences of the RR intervals (RMSSD) during 5 minutes after endotracheal intubation | 5 minutes after endotracheal intubation
  RMSSD represents the parasympathetic nervous activity mediated by a respiratory sinus arrhythmia.
Root mean square of the successive differences of the RR intervals (RMSSD) during 5 minutes before surgical incision | 5 minutes before surgical incision
  RMSSD represents the parasympathetic nervous activity mediated by a respiratory sinus arrhythmia.
Standard deviation of the RR intervals of normal sinus beats originating from the sinoatrial node of the right atrium (SDNN) during 5 minutes before anesthesia induction | 5 minutes before anesthesia induction
  SDNN represents the parasympathetic nervous activity mediated by a respiratory sinus arrhythmia.
Standard deviation of the RR intervals of normal sinus beats originating from the sinoatrial node of the right atrium (SDNN) during 5 minutes after anesthesia induction | 5 minutes after anesthesia induction
  SDNN represents the parasympathetic nervous activity mediated by a respiratory sinus arrhythmia.
Standard deviation of the RR intervals of normal sinus beats originating from the sinoatrial node of the right atrium (SDNN) during 5 minutes after endotracheal intubation | 5 minutes after endotracheal intubation
  SDNN represents the parasympathetic nervous activity mediated by a respiratory sinus arrhythmia.
Standard deviation of the RR intervals of normal sinus beats originating from the sinoatrial node of the right atrium (SDNN) during 5 minutes before surgical incision | 5 minutes before surgical incision
  SDNN represents the parasympathetic nervous activity mediated by a respiratory sinus arrhythmia.
The percentage of adjacent normal-to-normal sinus beat RR intervals that have a more than 50 milliseconds difference between them (pNN50) during 5 minutes before anesthesia induction | 5 minutes before anesthesia induction
  pNN50 represents the parasympathetic nervous activity mediated by a respiratory sinus arrhythmia.
The percentage of adjacent normal-to-normal sinus beat RR intervals that have a more than 50 milliseconds difference between them (pNN50) during 5 minutes after anesthesia induction | 5 minutes after anesthesia induction
  pNN50 represents the parasympathetic nervous activity mediated by a respiratory sinus arrhythmia.
The percentage of adjacent normal-to-normal sinus beat RR intervals that have a more than 50 milliseconds difference between them (pNN50) during 5 minutes after endotracheal intubation | 5 minutes after endotracheal intubation
  pNN50 represents the parasympathetic nervous activity mediated by a respiratory sinus arrhythmia.
The percentage of adjacent normal-to-normal sinus beat RR intervals that have a more than 50 milliseconds difference between them (pNN50) during 5 minutes before surgical incision | 5 minutes before surgical incision
  pNN50 represents the parasympathetic nervous activity mediated by a respiratory sinus arrhythmia.
Standard deviation 1 (SD1) of a Poincaré plot during 5 minutes before anesthesia induction | 5 minutes before anesthesia induction
  A Poincaré plot is a scatter plot where each pair of preceding and succeeding RR intervals is plotted on the abscissa and ordinate, respectively. After fitting the ellipse around the plot, SD1 is calculated as the standard deviation of the distance of each point from the line of identity (y=x). SD1 reflects the short-term HRV as the length of the transverse axis of the ellipse. SD1 correlates with the baroreflex sensitivity and HF.
Standard deviation 1 (SD1) of a Poincaré plot during 5 minutes after anesthesia induction | 5 minutes after anesthesia induction
  A Poincaré plot is a scatter plot where each pair of preceding and succeeding RR intervals is plotted on the abscissa and ordinate, respectively. After fitting the ellipse around the plot, SD1 is calculated as the standard deviation of the distance of each point from the line of identity (y=x). SD1 reflects the short-term HRV as the length of the transverse axis of the ellipse. SD1 correlates with the baroreflex sensitivity and HF.
Standard deviation 1 (SD1) of a Poincaré plot during 5 minutes after endotracheal intubation | 5 minutes after endotracheal intubation
  A Poincaré plot is a scatter plot where each pair of preceding and succeeding RR intervals is plotted on the abscissa and ordinate, respectively. After fitting the ellipse around the plot, SD1 is calculated as the standard deviation of the distance of each point from the line of identity (y=x). SD1 reflects the short-term HRV as the length of the transverse axis of the ellipse. SD1 correlates with the baroreflex sensitivity and HF.
Standard deviation 1 (SD1) of a Poincaré plot during 5 minutes before surgical incision | 5 minutes before surgical incision
  A Poincaré plot is a scatter plot where each pair of preceding and succeeding RR intervals is plotted on the abscissa and ordinate, respectively. After fitting the ellipse around the plot, SD1 is calculated as the standard deviation of the distance of each point from the line of identity (y=x). SD1 reflects the short-term HRV as the length of the transverse axis of the ellipse. SD1 correlates with the baroreflex sensitivity and HF.
Standard deviation 2 (SD2) of a Poincaré plot during 5 minutes before anesthesia induction | 5 minutes before anesthesia induction
  A Poincaré plot is a scatter plot where each pair of preceding and succeeding RR intervals is plotted on the abscissa and ordinate, respectively. After fitting the ellipse around the plot, SD2 is calculated as the standard deviation of the distance of each point from the line passing through the centroid, which vertically intersects the line of identity (y=x). SD2 reflects the long-term HRV as the length of the long axis of the ellipse. SD2 correlates with the baroreflex sensitivity and LF.
Standard deviation 2 (SD2) of a Poincaré plot during 5 minutes after anesthesia induction | 5 minutes after anesthesia induction
  A Poincaré plot is a scatter plot where each pair of preceding and succeeding RR intervals is plotted on the abscissa and ordinate, respectively. After fitting the ellipse around the plot, SD2 is calculated as the standard deviation of the distance of each point from the line passing through the centroid, which vertically intersects the line of identity (y=x). SD2 reflects the long-term HRV as the length of the long axis of the ellipse. SD2 correlates with the baroreflex sensitivity and LF.
Standard deviation 2 (SD2) of a Poincaré plot during 5 minutes after endotracheal intubation | 5 minutes after endotracheal intubation
  A Poincaré plot is a scatter plot where each pair of preceding and succeeding RR intervals is plotted on the abscissa and ordinate, respectively. After fitting the ellipse around the plot, SD2 is calculated as the standard deviation of the distance of each point from the line passing through the centroid, which vertically intersects the line of identity (y=x). SD2 reflects the long-term HRV as the length of the long axis of the ellipse. SD2 correlates with the baroreflex sensitivity and LF.
Standard deviation 2 (SD2) of a Poincaré plot during 5 minutes before surgical incision | 5 minutes before surgical incision
  A Poincaré plot is a scatter plot where each pair of preceding and succeeding RR intervals is plotted on the abscissa and ordinate, respectively. After fitting the ellipse around the plot, SD2 is calculated as the standard deviation of the distance of each point from the line passing through the centroid, which vertically intersects the line of identity (y=x). SD2 reflects the long-term HRV as the length of the long axis of the ellipse. SD2 correlates with the baroreflex sensitivity and LF.
Mean arterial blood pressure during 5 minutes before anesthesia induction | 5 minutes before anesthesia induction
  Measured at any time during 5 minutes before anesthesia induction
Mean arterial blood pressure during 5 minutes after anesthesia induction | 5 minutes after anesthesia induction
  Mean arterial blood pressure corresponding to the lowest systolic blood pressure during 5 minutes after anesthesia induction
Mean arterial blood pressure during 5 minutes after endotracheal intubation | 5 minutes after endotracheal intubation
  Measured at any time during 5 minutes after endotracheal intubation
Mean arterial blood pressure during 5 minutes before surgical incision | 5 minutes before surgical incision
  Measured at any time during 5 minutes before surgical incision
Systolic blood pressure during 5 minutes before anesthesia induction | 5 minutes before anesthesia induction
  Measured at any time during 5 minutes before anesthesia induction
Systolic blood pressure during 5 minutes after anesthesia induction | 5 minutes after anesthesia induction
  The lowest systolic blood pressure during 5 minutes after anesthesia induction
Systolic blood pressure during 5 minutes after endotracheal intubation | 5 minutes after endotracheal intubation
  Measured at any time during 5 minutes after endotracheal intubation
Systolic blood pressure during 5 minutes before surgical incision | 5 minutes before surgical incision
  Measured at any time during 5 minutes before surgical incision
Bispectral index (BIS) during 5 minutes before anesthesia induction | 5 minutes before anesthesia induction
  The BIS value corresponding to blood pressure measured during 5 minutes before anesthesia induction
Bispectral index (BIS) during 5 minutes after anesthesia induction | 5 minutes after anesthesia induction
  The BIS value corresponding to the lowest systolic blood pressure during 5 minutes after anesthesia induction
Bispectral index (BIS) during 5 minutes after endotracheal intubation | 5 minutes after anesthesia induction
  The BIS value corresponding to blood pressure measured during 5 minutes after endotracheal intubation
Bispectral index (BIS) during 5 minutes before surgical incision | 5 minutes before surgical incision
  The BIS value corresponding to blood pressure measured during 5 minutes before surgical incision

OTHER OUTCOMES:
Deceleration capacity (DC) during 5 minutes before anesthesia induction | 5 minutes before anesthesia induction
  The quasi-periodic decelerations in short-term heart rate are calculated using a phase-rectified signal averaging technique. The calculated deceleration (deceleration capacity: DC) represents parasympathetic nervous activity.
Deceleration capacity (DC) during 5 minutes after anesthesia induction | 5 minutes after anesthesia induction
  The quasi-periodic decelerations in short-term heart rate are calculated using a phase-rectified signal averaging technique. The calculated deceleration (deceleration capacity: DC) represents parasympathetic nervous activity.
Deceleration capacity (DC) during 5 minutes after endotracheal intubation | 5 minutes after endotracheal intubation
  The quasi-periodic decelerations in short-term heart rate are calculated using a phase-rectified signal averaging technique. The calculated deceleration (deceleration capacity: DC) represents parasympathetic nervous activity.
Deceleration capacity (DC) during 5 minutes before surgical incision | 5 minutes before surgical incision
  The quasi-periodic decelerations in short-term heart rate are calculated using a phase-rectified signal averaging technique. The calculated deceleration (deceleration capacity: DC) represents parasympathetic nervous activity.
Diastolic blood pressure during 5 minutes before anesthesia induction | 5 minutes before anesthesia induction
  Measured at any time during 5 minutes before anesthesia induction
Diastolic blood pressure during 5 minutes after anesthesia induction | 5 minutes after anesthesia induction
  Diastolic blood pressure corresponding to the lowest systolic blood pressure during 5 minutes after anesthesia induction
Diastolic blood pressure during 5 minutes after endotracheal intubation | 5 minutes after endotracheal intubation
  Measured at any time during 5 minutes after endotracheal intubation
Diastolic blood pressure during 5 minutes before surgical incision | 5 minutes before surgical incision
  Measured at any time during 5 minutes before surgical incision

CONTACTS AND LOCATIONS:
Overall Officials: Jonghae Kim, M.D., Principal Investigator — Daegu Catholic University Medical Center
Locations (1):
- Daegu Catholic University Medical Center, Daegu, South Korea